CLINICAL TRIAL: NCT05576701
Title: The Effect of Laughter Therapy on Acceptance of Disease, Adherence to Treatment and Comfort Level in Patients Receiving Hemodialysis Treatment: A Randomized Controlled Trial
Brief Title: Laughter Therapy Application in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bozok University (Other)
Responsible Party: Principal Investigator, Betül Bal, Lecturer, Bozok University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BBal
Record Dates: First submitted 2022-09-10; First posted 2022-10-12 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Comfort; Acceptance Processes; Hemolysis; Laughter Therapy; Treatment Adherence; Patients
MeSH Terms: conditions — Behavior; Hemolysis; Treatment Adherence and Compliance | interventions — Laughter Therapy

STUDY DESIGN:
Intervention Model Description: While the patients were randomized; In order to keep the possibility of being affected by each other at a minimum level, the work was continued with the same application group in the same session group. 72 days in universe, hemodialysis days and sessions at time of day, next Wednesday, Friday = 36 patients); Tuesday, Thursday, evening patient control (n=36 patients are guided by the drawing method.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laughter Therapy (Experimental): Laughter therapy consists of group-based interventions that include yoga breathing exercises and stillness. Laughter education is a form of exercise with gratuitous laughter and childlike play. Laughter therapy practices consist of four steps. These; warming exercises, deep exercises, playing childlike games and entertainment (eg greeting laughter, lion laughter, milk waving sounds, quiet laughter, etc.). Laughter therapy sessions in the study were carried out for 4 weeks and three times a week. Laughter therapy has been applied by researchers who have a leader certificate.
  Interventions: Behavioral: Laughter Therapy
- Control (Active Comparator): The patients in the control group, on the other hand, did not undergo any intervention other than their routine treatment and care. The patients were followed for four weeks. Before the study, data collection tools were applied to the patients. Again, after the study started and the study ended, all other data collection tools were applied, except the "Patient Information Form".
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Laughter Therapy — In this study, laughter therapy was applied to the experimental group three times a week (on Mondays, Wednesdays, and Fridays) for a total of 12 sessions. Each session started with other patients in the HD unit while the patient was receiving HD treatment (1 hour after HD started) and lasted 30-45 minutes. The number of patients who will take part in each laughter session is based on the number of patients attending that session in the hemodialysis unit.
  Arms: Laughter Therapy
Other: Control — The patients in the control group, on the other hand, did not undergo any intervention other than their routine treatment and care. Laughter therapy was applied for four weeks to HD patients in the control group who wanted the results of the research.
  Arms: Control

SUMMARY:
Background: A randomized controlled study was conducted on the effects of laughter therapy on increasing the acceptance of the disease, compliance with treatment and comfort levels in patients receiving hemodialysis treatment.

Materials and methods: The study was conducted with 42 (experimental group=21, control group=21) patients treated in the hemodialysis unit. Eight sessions of laughter yoga were applied to the hemodialysis patients in the experimental group for four weeks, two days a week. Data were used on the Patient Information Form, the Acceptance Scale, the End Stage Renal Failure - Compliance Scale, and the Hemodialysis Comfort Scale.

DETAILED DESCRIPTION:
Kidney Failure is an important public health problem due to its increasing prevalence and high costs worldwide. Especially patients in the end stage of renal failure (ESRD) are faced with a life-threatening chronic disease. These patients need lifelong treatment and care to minimize the negative effects of impaired kidney function and to maintain life.

In the treatment and recovery processes of chronic diseases such as kidney failure, individuals' acceptance of the disease, compliance with the treatment and their comfort level are very important. The stage of acceptance of the disease is when the individual learns to live with the chronic disease by adapting to various complications and changes related to the chronic disease. Not accepting the disease results in submission to the problems brought about by the disease and causes an increase in the sense of dependency and a decrease in the sense of self-efficacy and self-esteem. It is very difficult for patients with end-stage renal disease who receive hemodialysis (HD) treatment among chronic diseases to accept the disease because they are affected by many physical, mental, spiritual and social aspects. It has been reported that patients receiving HD treatment often experience problems in the acceptance process of the disease. In the literature, it has been emphasized that acceptance of the disease is effective in reducing the physical, psychosocial and emotional problems caused by HD treatment. In addition, it has been shown that accepting the disease is effective in increasing the quality of life by reducing symptoms such as fatigue, constipation, loss of appetite, sexual dysfunction and stress in HD patients. On the other hand, it has been determined that individuals with low acceptance level of the disease have increased complaints about the disease and treatment. In studies related to the subject, it has been determined that patients' acceptance of the disease is at different levels.

Another important step in the treatment and recovery processes of chronic diseases is compliance with treatment. Compliance with treatment in the management of HD disease greatly affects the success of treatment. Compliance with treatment in HD patients; It is considered as compliance with fluid-diet-drug intake and participation in hemodialysis sessions. In studies, 55-77% of individuals receiving HD treatment have fluid restriction 30-70% diet restriction, 38-75% of drug intake and participation in 30-69% HD sessions have been found to have problems with it. This situation increases hospitalization, morbidity and mortality rates in individuals receiving HD treatment and creates a heavy burden on the health system. Therefore, it is important to increase patients' acceptance of the disease and their compliance with treatment.

Many physical and psychosocial symptoms occur during the disease and treatment processes, and the care needs of individuals who experience physical, social, economic and psychological problems increase, and there is a significant decrease in the quality of life and comfort. Helping patients with their needs, providing peace and being able to overcome problems gain priority. Therefore, the comfort that defines this situation; plays an important role in the care of individuals with chronic diseases. Comfort; It is defined as meeting the needs of individuals, solving their problems, reaching the desired result and peace by considering them as a whole in terms of physical, psychological, social and environmental aspects. Today, many complications and unmet basic needs of individuals with chronic diseases affect their comfort levels negatively. In the studies conducted, the comfort level of individuals receiving HD treatment is low and moderate. In the literature, problems such as painful invasive procedures, fatigue, decrease in energy, itching, bone/joint pain, numbness or tingling in the feet, sleep problems, dry mouth, decreased sexual desire and arousal experienced by individuals who receive HD treatment can lower their comfort levels. negatively. In order for patients to cope with the problems related to HD treatment, the level of comfort needs to be increased.

It is seen that some complementary methods are used in the literature to increase the health level of patients receiving HD treatment and to ensure that they can lead a quality life. One of these methods is laughter therapy. Laughter therapy; Developed in India in 1995, yoga is a group-based initiative that includes breathing exercises and simulated laughter. It is also a type of exercise done by singing songs, laughing for no reason and playing childish games. Laughter therapy for cardiovascular disease; irritable bowel syndrome, chronic obstructive pulmonary disease, diabetes, cancer. It has been dealt with many diseases such as and Parkinson's and it has been found to have beneficial effects on these diseases. In a randomized controlled experimental study conducted by Bennet et al. in patients receiving HD treatment, it was found that laughter therapy reduced the symptoms of depression. In the study of Sousa et al., it was determined that laughter therapy increases subjective happiness and significantly reduces symptoms of depression. In other studies conducted in patients receiving HD treatment, laughter therapy has positive effects on anxiety, depression, stress, and happiness was determined. There are also studies that show that laughter therapy regulates blood pressure in patients receiving HD treatment. In all these studies, it was observed that laughter therapy is a safe and feasible intervention in patients receiving HD treatment. When the literature is examined, no studies have been found on the effects of laughter therapy on the acceptance of the disease, compliance with the treatment and comfort level, although complementary methods are frequently used in studies on patients. In this direction, it was aimed to evaluate the effects of laughter therapy on acceptance of the disease, compliance with treatment and comfort levels in patients receiving HD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated for HD for more than six months,
* who are over 18 years old
* who agree to participate in the study

Exclusion Criteria:

* patients with severe cardiovascular disease,
* who are pregnant,
* with psychiatric disorders,
* who do not regularly attend laughter therapy sessions,
* who have experience in laughter therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Change in Disease Acceptance Level | 4 weeks
  This form was used to measure the degree of acceptance of the disease in hemodialysis patients. In the research, it was applied twice in total before the laughter therapy was applied and after the laughter therapy was finished. The total score to be obtained from the scale varies between 8 and 40, and as the score increases, the level of acceptance of the disease increases.

SECONDARY OUTCOMES:
Change in compliance level in end-stage renal disease | 4 weeks
  This form was used to evaluate participation in hemodialysis, medication adherence, fluid compliance, and diet compliance in hemodialysis patients. In the research, it was applied twice in total before the laughter therapy was applied and after the laughter therapy was finished. The range of scores that can be obtained from the scale is between 0-1200, and as the score increases, the compliance of the patients with the treatment also increases.

OTHER OUTCOMES:
Change in comfort level in hemodialysis patients | 4 weeks
  This form was used to evaluate the comfort levels of individuals who received hemodialysis treatment for at least 6 months. In the research, it was applied twice in total before the laughter therapy was applied and after the laughter therapy was finished.The lowest score that can be obtained from the scale is 9, and the highest is 45. As the score gets closer to 45, the comfort level increases.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Betül, Yozgat, Akdağmadeni
  - Betül, Yozgat